CLINICAL TRIAL: NCT05275088
Title: An Exploratory Study to Evaluate the Prizvalve® System in Patients With Severe Atrioventricular Annular Calcification or Failed Prosthetic Atrioventricular Valve/ Annulus Repair
Brief Title: Prizvalve® Transcatheter Atrioventricular Valve Replacement Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai NewMed Medical Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-valve-2021-12
Record Dates: First submitted 2022-02-25; First posted 2022-03-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Atrioventricular Annular Calcification; Failed Prosthetic Atrioventricular Valve/ Annulus Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Transcatheter atrioventricular valve replacement with the Prizvalve® system
  Interventions: Device: Prizvalve® system

INTERVENTIONS:
Device: Prizvalve® system — Transcatheter atrioventricular valve replacement

SUMMARY:
To evaluate the safety and performance of the Prizvalve® system in patients with severe atrioventricular annular calcification or failed prosthetic atrioventricular valve/ annulus repair.

DETAILED DESCRIPTION:
The Prizvalve® study is a single-center, single-arm, prospective, exploratory clinical study.

ELIGIBILITY:
1. Inclusion criteria for patients with severe atrioventricular valve annular calcification:

1. Atrioventricular valve annular calcification with moderate or severe atrioventricular valve disease (stenosis, regurgitation, or mixed);
2. Patient with symptoms, and NYHA Functional Class≥Ⅱ;
3. 18 years and older who is not in pregnancy or lactation;
4. Life expectancy>12 months;
5. Patient who is anatomically suitable for transcatheter atrioventricular valve replacement;
6. According to the evaluation of the heart team, the patient can benefit from transcatheter atrioventricular valve replacement;
7. The patient can understand the purpose of the trial, voluntarily participate in and sign the informed consent form, and is willing to accept relevant examinations and clinical follow-ups;
8. Patient with high risk of routine surgery (STS>8%) or severe comorbidities that is not suitable for surgery, or with severely calcified valve annulus that cannot be operated.

2. Inclusion criteria for patients with failed prosthetic atrioventricular valve/annulus repair:

1. The patient has undergone atrioventricular valve replacement or valve annulus repair in the past, accompanied by severe atrioventricular valve regurgitation or stenosis;
2. The patient is symptomatic with NYHA Functional Class≥II or hemolytic anemia requiring blood transfusion (no other causes of hemolytic anemia were found after examination);
3. 18 years and older who is not in pregnancy or lactation;
4. Patient who is anatomically suitable for transcatheter atrioventricular valve replacement;
5. According to the evaluation of the heart team, the patient can benefit from transcatheter atrioventricular valve replacement;
6. The patient can understand the purpose of the trial, voluntarily participate in and sign the informed consent form, and is willing to accept relevant examinations and clinical follow-ups;
7. Patient with high risk of routine surgery (STS>8%) or severe comorbidities that is not suitable for surgery.

Exclusion criteria:

1. Evidence of an acute myocardial infarction <1 month(30 days) before the intended treatment;
2. Any therapeutic cardiac operation (excluding previous PCI and pacemaker implantation) is performed within 30 days of the index procedure;
3. Patient with planned concomitant surgical or transcatheter ablation for atrial fibrillation;
4. Patient with hypertrophic cardiomyopathy with obstruction;
5. Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) <20%;
6. Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
7. Acute peptic ulcer or upper gastrointestinal bleeding within 3 months prior to procedure;
8. Allergy to cobalt-chromium alloy or contrast agent; inability to tolerate anticoagulation and antiplatelet therapy;
9. Active stage of infective endocarditis or other active infection;
10. Cerebrovascular accident within 3 months prior to procedure, excluding transient ischemic attack;
11. Patient with poor compliance and could not complete the study as required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2028-06-10 (Estimated)

PRIMARY OUTCOMES:
Technical success | 30 days
  Definition:
  1. Freedom from death;
  2. Successful vascular delivery and retrieval of transcatheter valve delivery system;
  3. Correct position of transcatheter valve;
  4. No need for any emergency surgery or re-intervention (including device-related and surgical approach-related);
  5. Adequate performance of prosthesis (mean pressure gradient (MVG) <10mmHg, valve regurgitation <2+).

SECONDARY OUTCOMES:
Procedural Success | 30 days,1 year
  1. Device success;
  2. No SAE's including: death; stroke; life threatening bleeding; major vascular complications; secondary severe cardiac organic disease (eg: aortic dissection, apical aneurysm formation, left ventricular outflow tract obstruction, etc.); stage 2 or 3 AKI; MI or coronary ischemia requiring PCI or CABG; severe hypotension; heart failure or respiratory failure requiring high-dose vasoactive drugs/or cardiac mechanical assist devices; any valve-related dysfunction including migration, thrombosis, or other complication requiring surgery or repeat intervention.
Device success | 30 days,1 year
  Definitions:
  1. Freedom from stroke;
  2. Prosthetic heart valve function is normal (including no displacement, calcification, thrombosis, hemolysis, or endocarditis);
  3. No need for any emergency surgery or secondary intervention (including device-related and surgical approach-related);
  4. No atrioventricular valve stenosis (mean pressure gradient <10mmHg);
  5. Atrioventricular valve regurgitation <2+ (including central leakage and paravalvular leakage), and no related hemolysis;
  6. LVOT pressure gradient increased <20mmHg.
All-cause mortality | 30 days,1 year
  All-cause mortality included cardiac and non-cardiac death.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China